CLINICAL TRIAL: NCT04697290
Title: A Study of CD19/CD20 Dual CAR-T Cells in the Treatment of Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma(B-NHL)
Brief Title: CD19/CD20 Dual-CAR-T in B-cell Non-Hodgkin's Lymphoma Patients.
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Plan adjustment
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: China Immunotech Pharmaceuticals Co.Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-012
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD20 Dual-CAR-T cells (Experimental): CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest for at least 2 days before infusion.
  Interventions: Biological: CD19/CD20 Dual-CAR-T cells

INTERVENTIONS:
Biological: CD19/CD20 Dual-CAR-T cells — CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest at least for 2 days before infusion. CD19/CD20 Dual-CAR-T cells will be intravenously infused with a escalated dose of 2E6、6E6、1E7、3E7 cells/kg.

SUMMARY:
This is a single center, single arm, open-label, phase I study to evaluate the safety and efficacy of CD19/CD20 Dual-CAR-T cells in patients with refractory or relapsed B-NHL.

DETAILED DESCRIPTION:
This Phase I study is designed as a pilot trial evaluating the safety and efficacy of CD19/CD20 Dual-CAR-T cell therapy in subjects with refractory and relapsed B-NHL. Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of CD19/CD20 Dual-CAR-T cells. Safety and efficacy of CD19/CD20 Dual-CAR-T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19/CD20 Dual-CAR-T cells therapy in patients with refractory and relapsed B-NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. NHL confirmed by cytology or histology, including diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, etc.
3. Relapse or refractory after at least second-line treatment;
4. With evaluable target lesions.Measurable target lesions: lymph nodes>1.5x1.0cm, extranodal lesions>1.0x1.0cm;
5. Double positive expression of CD19 / CD20 in B cells;
6. ECOG score 0-2 points;
7. Good organ function:

   Blood routine: absolute neutrophil count (ANC) ≥1.0×109/L; hemoglobin (Hb) ≥80 g/L; platelet count (PLT) ≥50×109/L; Blood biochemistry: total bilirubin≤3×upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤3×upper limit of normal (ULN); Pulmonary function: ≤CTCAE Grade 1 dyspnea and SaO2≥92% in indoor air environment; Heart function: Left ventricular ejection fraction (LVEF) ≥50%.
8. Women of childbearing age (15-49 years old) must receive a pregnancy test within 7 days prior to initiation of treatment and the results are negative; male and female patients with fertility must use an effective contraceptive to ensure 3 months after discontinuation of treatment during the study period not pregnant inside;
9. Patients who voluntarily sign informed consent and are willing to comply with treatment plans.

Exclusion Criteria:

1. Active infections that are difficult to control;
2. Active hepatitis B, active hepatitis C, human immunodeficiency virus (HIV) antibody positive, and Treponema pallidum antibody test positive;
3. The tumor invades the central nervous system or primary CNS lymphoma;
4. Anti-GVHD (acute or chronic) treatment is being performed within 4 weeks before apheresis and cell infusion;
5. Have undergone the following treatments:

   * Those who have received chemotherapy or radiotherapy 5 days before apheresis;
   * Those who have used drugs that stimulate the production of bone marrow hematopoietic cells within 5 days before apheresis;
   * Received donor lymphocyte infusion (DLI) within 6 weeks before cell infusion;
   * Have received autologous hematopoietic stem cell transplantation (HSCT) 3 months before apheresis, or received allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 12 months;
   * Have used any gene therapy products before;
6. History of epilepsy or other central nervous system diseases; or clinically diagnosed as having severe thyroid dysfunction; or active autoimmune diseases;
7. History of other malignant tumors that have not been remission for at least 3 years ;
8. Any of the following cardiovascular diseases occurred within 6 months of the screening period, including NYHA heart function grade III or IV heart failure, cardiovascular angioplasty or stent, myocardial infarction, unstable angina, or other clinical symptoms Significant heart disease;
9. Pregnant or lactating women;
10. The investigator believes that there are other factors that are not suitable for selection or that affect subjects' participation or completion of the study.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 6months
  Percentage of participants with adverse events.
Objective remission rate(ORR) | 6 months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants.

SECONDARY OUTCOMES:
Relapse-Free Survival(RFS ) | 6 months
Overall-Survival(OS) | 6 months

OTHER OUTCOMES:
Persistence of CAR-T cells in vivo | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China